CLINICAL TRIAL: NCT03920501
Title: Comparison of Tele-Critical Care Versus Usual Care On ICU Performance: A Cluster Randomized Clinical Trial
Brief Title: Comparison of Tele-Critical Care Versus Usual Care On ICU Performance (TELESCOPE)
Acronym: TELESCOPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TELESCOPE
Record Dates: First submitted 2019-04-10; First posted 2019-04-19 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-08

CONDITIONS: Critical Care; Intensive Care Unit
Keywords: Critical care; Quality improvement; Tele-critical care; Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-Critical Care (Experimental): Tele-Critical Care + Audit & Feedback.
  Interventions: Behavioral: Tele-Critical Care
- Usual Care (No Intervention): Usual Care.

INTERVENTIONS:
Behavioral: Tele-Critical Care — Daily multidisciplinary rounds with a board certified physician through tele-critical care focusing on: 1) diagnosis; 2) active problems; and 3) therapeutic goals. In addition, the management of health care quality indicators will be conducted by a specially trained (Science of Improvement) board-certified intensive care physician.
  Arms: Tele-Critical Care

SUMMARY:
TELESCOPE will be a cluster randomized clinical trial to ascertain whether the use of an intervention including multidisciplinary round with a board certified physician through tele-critical care and periodic meetings to discuss strategies to improve quality indicators can reduce ICU length of stay of patients admitted to intensive care units (ICUs).

DETAILED DESCRIPTION:
Cluster randomized trial involving ICUs in Brazil. ICU is the unit of randomization.

The trial will have two stages:

Stage I - Baseline data:

* Characterize participant ICUs and quality indicators
* Characterize patients from each participant ICU to describe baseline outcomes

Stage II - Intervention:

This is the main stage for data analysis. ICUs will be randomly assigned to an experimental or control group. The experimental group should use a multidisciplinary rounds with a board certified physician through tele-critical care and take part in meetings to discuss how to improve local quality indicators, and the control group will follow the local standard of care.

ELIGIBILITY:
Inclusion Criteria for Clusters:

* Intensive care units from public hospitals and with at least eight beds
* Intensive care units with physician and nurses available 24 hours a day

Exclusion Criteria for Clusters:

* Intensive care units with structured multidisciplinary round more than three times a week based in a formal instrument
* Intensive care units already doing audit & feedback
* Dedicated coronary care units/cardiac intensive care units or other specialized units
* Step-down units

Inclusion Criteria for Patients:

* Adult patients (> 18 years old)
* Admitted after the beginning of the study

Exclusion Criteria for Patients:

* Admission for other reasons than medical (e.g., judicial cause)
* Previously included in TELESCOPE (for the primary outcome analysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19360 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Intensive Care Unit Length of Stay | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Time until discharge from the intensive care unit

SECONDARY OUTCOMES:
In-Hospital Mortality | From date of randomization until the date of hospital discharge or death, whichever comes first, assessed up to 90 days
  Any death during hospital stay
Standardized Resource Use | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Calculated based on length of stay in the intensive care unit and adjusted for severity of acute illness
Standardized Mortality Rate | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Ratio of observed deaths to expected deaths
Incidence Density of Central Line-Associated Bloodstream Infection (CLABSI) | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Following the Centers for Disease Control/National Healthcare Safety Network (CDC/NHSN) Surveillance Definition of Healthcare-Associated Infection 2019
Incidence Density of Ventilator-Associated Pneumonia (VAP) | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Following the Centers for Disease Control/National Healthcare Safety Network (CDC/NHSN) Surveillance Definition of Healthcare-Associated Infection 2019
Incidence Density of Urinary Tract Infection Associated with Catheter | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Following the Centers for Disease Control/National Healthcare Safety Network (CDC/NHSN) Surveillance Definition of Healthcare-Associated Infection 2019
Ventilator-Free Days at Day 28 | 28 Days
  Survival time free of invasive mechanical ventilation from ICU admission to day 28.
Patient-Days Receiving Oral or Enteral Feeding | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Use of enteral or oral feeding
Patient-Days Under Light Sedation or Alert and Calm | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Defined as a Richmond Agitation-Sedation Scale (RASS) -3 to +1
Rate of Patients Under Normoxia | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Defined as oxygen saturation (SpO2) between 92% and 96%

OTHER OUTCOMES:
Rate of Patients with Head of the Bed Elevated | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  30 degrees in patients under mechanical ventilation
Incidence of Early Reintubation | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Less than 48 hours after extubation
Incidence of Accidental Extubation | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Rate of accidental extubation
Rate of Central-Line Catheter Use | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Use of central-line catheter use
Rate of Vesical Catheter Use | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Use of vesical catheter
Rate of Adequate Prophylaxis for Venous Thromboembolism | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Adequate prophylaxis for venous thromboembolism
Rate of Adequate Glycemic Control | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  Adequate glycemic control
ICU Readmission | From date of randomization until the date of hospital discharge or death, whichever comes first, assessed up to 90 days
  Readmission less than 24 hours after discharge
ICU Mortality | From date of randomization until the date of ICU discharge or death, whichever comes first, assessed up to 90 days
  ICU mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Adriano J Pereira, MD PhD, Study Director — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data sharing open to researchers not members of the study after two years of the publication of the main study
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: After two years of the first publication
Access Criteria: Data will be acessed through an online repository protected with password and for secondary analyses according to pre-specified plans.

REFERENCES:
- [Derived] Pereira AJ, Noritomi DT, Dos Santos MC, Correa TD, Ferraz LJR, Schettino GPP, Cordioli E, Morbeck RA, Morais LC, Salluh JIF, Azevedo LCP, Biondi RS, Rosa RG, Cavalcanti AB, Berwanger O, Serpa Neto A, Ranzani OT. Effect of Tele-ICU on Clinical Outcomes of Critically Ill Patients: The TELESCOPE Randomized Clinical Trial. JAMA. 2024 Dec 3;332(21):1798-1807. doi: 10.1001/jama.2024.20651. PMID 39382244
- [Derived] Ranzani O, Pereira AJ, Santos MCD, Correa TD, Ferraz LJR, Cordioli E, Morbeck RA, Berwanger O, Morais LC, Schettino G, Cavalcanti AB, Rosa RG, Biondi RS, Salluh JIF, Azevedo LCP, Serpa Neto A, Noritomi DT. Statistical analysis of a cluster-randomized clinical trial on adult general intensive care units in Brazil: TELE-critical care verSus usual Care On ICU PErformance (TELESCOPE) trial. Rev Bras Ter Intensiva. 2022 Jan-Mar;34(1):87-95. doi: 10.5935/0103-507x.20220003-pt. PMID 35766658
- [Derived] Noritomi DT, Ranzani OT, Ferraz LJR, Dos Santos MC, Cordioli E, Albaladejo R, Serpa Neto A, Correa TD, Berwanger O, de Morais LC, Schettino G, Cavalcanti AB, Rosa RG, Biondi RS, Salluh JI, Azevedo LCP, Pereira AJ; TELESCOPE Trial Investigators. TELE-critical Care verSus usual Care On ICU PErformance (TELESCOPE): protocol for a cluster-randomised clinical trial on adult general ICUs in Brazil. BMJ Open. 2021 Jun 21;11(6):e042302. doi: 10.1136/bmjopen-2020-042302. PMID 34155070

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT03920501/SAP_000.pdf